CLINICAL TRIAL: NCT01652235
Title: Study Assessing Safety and Effectiveness of Perivisceral Aortic Aneurysm Treatment With the Zenith® Fenestrated AAA Endovascular Graft and the Zenith® p-Branch® and the Effects on Organ and Extremity Perfusion
Brief Title: Zenith® p-Branch® and Zenith® Fenestrated AAA Endovascular Graft Clinical Study
Acronym: FENP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-003
Record Dates: First submitted 2012-07-17; First posted 2012-07-30 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Abdominal aortic aneurysm; Endovascular; Fenestration; Juxtarenal; Off-the-shelf; Pararenal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endovascular (Experimental): Zenith® p-Branch® or Zenith® Fenestrated AAA Endovascular Graft
  Interventions: Device: Zenith® p-Branch® or Zenith® Fenestrated AAA Endovascular Graft

INTERVENTIONS:
Device: Zenith® p-Branch® or Zenith® Fenestrated AAA Endovascular Graft — Instead of making a large incision in the chest, the physician makes a small incision near each hip to insert, and guides the study device(s) into place in the aorta.
  Other Names: Endovascular stent; Stent-graft

SUMMARY:
The Zenith® p-Branch® and Zenith® Fenestrated AAA Endovascular Graft Single-Center Study is a clinical trial approved by US FDA to study the safety and effectiveness of the Zenith® p-Branch® and Zenith® Fenestrated AAA Endovascular Graft in the treatment of abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal aortic aneurysm > 5.0 cm or 2 times the normal aortic diameter
* Abdominal aortic aneurysm with history of growth > 0.5 cm in 6 months
* Penetrating juxtarenal aortic ulcer > 10 mm in depth and 20 mm in diameter

Exclusion Criteria:

* Age < 18 years
* Life expectancy < 2 years
* Pregnant or breast feeding
* Inability or refusal to give informed consent
* Unwilling or unable to comply with the follow-up schedule
* Additional medical restrictions as specified in the Clinical Investigation Plan
* Additional anatomical restrictions as specified in the Clinical Investigation Plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-07; Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. McKinsey, MD, Principal Investigator — Mount Sinai-West
Locations (2):
- United States (2):
  - Mount Sinai-West, New York, New York
  - New York Presbyterian Hospital System, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Endovascular: Experimental: Endovascular
  Zenith® p-Branch® or Zenith® Fenestrated AAA Endovascular Graft
Period: Overall Study
Arm/Group | Endovascular
Started | 28
Completed | 12
Not Completed | 16
Not completed — Death | 9
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 22
Age, Continuous [Mean (Full Range); unit: Years] | 73.2 [59 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24
  Hispanic or Latino | 2
  Black or African American | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Technical Success:
Description: Successful access of the aneurysm site and deployment of the Zenith® Fenestrated AAA Endovascular Graft or the Zenith® p-Branch™ in the intended location. The endovascular graft and all vessels targeted with fenestrations must be patent at the time of deployment completion as evidenced by intraoperative angiography
Time Frame: Immediately post graft deployment
Measure: Number; unit: participants
Arm/Group | Endovascular
Number analyzed (Participants) | 28
participants | 28

2. Primary Outcome: Procedural Success
Description: Technical Success, with all of the following at post-procedure (within 30 days):
  * No type I or type III endoleaks;
  * No procedure related serious adverse events or major complications;
  * Patency of the endovascular graft and all vessels targeted with fenestrations as evidenced by CT scan, angiography or by duplex ultrasound in those patients experiencing renal failure or otherwise unable to undergo contrast enhanced CT scan.
Time Frame: Within 30 days post graft deployment
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular
Number analyzed (Participants) | 28
Participants | 25

3. Primary Outcome: Treatment Success
Description: Procedural Success, with all of the following at 12 months:
  * No type I or type III endoleaks;
  * No serious adverse events or major complications;
  * No aneurysm enlargement greater than 0.5 cm;
  * Patency of the endovascular graft and all vessels targeted with fenestrations as evidenced by CT scan, angiography or by duplex ultrasound in those patients experiencing renal failure or otherwise unable to undergo contrast enhanced CT scan.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular
Number analyzed (Participants) | 28
Participants | 23

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Endovascular
All-Cause Mortality (participants affected / at risk) | 9/28
Serious Adverse Events (participants affected / at risk) | 4/28
Other Adverse Events (participants affected / at risk) | 20/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular (N=28)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular (N=28)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (4)
Blood creatinine increased (Investigations) | 7 (8)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Renal artery occlusion (Renal and urinary disorders) | 3 (3)
Renal infarct (Renal and urinary disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Mechanical ventilation (Surgical and medical procedures) | 2 (2)
Oxygen therapy (Surgical and medical procedures) | 2 (2)
Transfusion (Surgical and medical procedures) | 8 (9)
Aneurysm (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT01652235/Prot_000.pdf